CLINICAL TRIAL: NCT00799539
Title: An International Single-Arm Study to Provide Further Safety and Efficacy Data on the Bortezomib(Velcade)/Melphalan/Prednisone Regimen in Previously Untreated Transplant Ineligible Multiple Myeloma Patients
Brief Title: A Study to Further Assess Safety and Effectiveness Data of the Bortezomib(Velcade)/Melphalan/Prednisone (BMP) Regimen in Previously Untreated and Transplant Ineligible Multiple Myeloma Patients
Status: No longer available | Type: Expanded Access
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Collaborators: Ortho Biotech Canada (Unknown)
Responsible Party: Sponsor
Other Study IDs: CR015310; 26866138MMY3020 (Other: Janssen-Ortho, Canada)
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Myeloma
Keywords: Prednisone; Bortezomib; Melphalan
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone

INTERVENTIONS:
Drug: bortezomib — From cycles 1-4, 1.3mg/m^2 on days 1,4,8,11,22,25,29,and 32 of each 6-week cycle
Drug: bortezomib — From cycles 5-9, 1.3mg/m^2 on days 1, 8, 22, and 29 of each 6-week cycle
Drug: melphalan — 9 mg/m^2 once daily on days 1-4 of each 6-week cycle
Drug: prednisone — 60 mg/m^2 once daily on days 1-4 of each 6-week cycle

SUMMARY:
The primary reason for this study is to further assess safety and efficacy data of the bortezomib/melphalan/prednisone (BMP) regimen in previously untreated and transplant ineligible multiple myeloma patients

DETAILED DESCRIPTION:
OBJECTIVES: The primary objective of this study is to further assess safety and efficacy data of the bortezomib/melphalan/prednisone (BMP) regimen in previously untreated and transplant ineligible multiple myeloma patients. This is an international, multicentred, open-label, single-arm, non-comparative study. After providing written informed consent, patients will be evaluated for eligibility during a screening period of 14 days (Days -14 to Day -1). Baseline efficacy and safety assessments will be performed on Day 1 (the first day of treatment) prior to the study drug administration for patients with measurable monoclonal paraprotein (M-protein) or within at least 14 days for patients with extramedullary plasmacytomas. Patients with previously untreated multiple myeloma who are not candidates for high dose chemotherapy with stem cell transplant high dose therapy/stem cell transplant (HDT/SCT) will be enrolled. Approximately 150 patients will be enrolled on study. Patients will receive BMP treatment, consisting of Bortezomib (twice weekly [Days 1, 4, 8, 11, 22, 25, 29 and 32] for four 6-week cycles [8 doses per cycle] followed by once weekly [Days 1, 8, 22, and 29] for five 6-week cycles [4 doses per cycle]) in combination with melphalan and prednisone once daily on Days 1 to 4 of each 6-week cycle. Treatment will continue for a maximum of 9 cycles (54 weeks) and will be discontinued if disease progression or an unacceptable treatment-related toxicity occurs, or if a patient withdraws consent. The Final Visit/Early Termination Visit will occur 30-42 days after the last dose of Bortezomib. Investigators will be asked to report on TTP every 6 months from Final Visit until disease progression for a period of up to 2 years. Safety will be assessed by the monitoring of adverse events, physical (including neurological/peripheral neurological) examinations, vital sign measurements, hematology and clinical chemistry tests. Karnofsky performance status and FACT/GOG-Ntx will also be assessed. Efficacy evaluations of serum and urine M-protein levels together with extramedullary plasmacytoma evaluations will be done at the beginning of each cycle. Investigator reported TTP and subsequent therapy will also be captured.

The secondary objectives are to assess neurotoxicity using the FACT/GOG-Ntx questionnaire, and to capture investigator reported time to progression (TTP) data. STUDY POPULATION: The patient population comprises a maximum of 150 male and female patients, who have symptomatic multiple myeloma or asymptomatic multiple myeloma with related organ or tissue damage, presence of measurable disease, Karnofsky performance status score greater than or equal to 60 points, and clinical hematology and chemistry laboratory values that meet predefined criteria. It is expected that approximately 150 patients will be enrolled. Potential patients will be excluded who are candidates for HDT/SCT; have a diagnosis of smoldering multiple myeloma, monoclonal gammopathy of undetermined significance (MGUS), or Waldenström's disease; have had prior or current systemic therapy for multiple myeloma; have had radiation therapy, plasmapheresis, or major surgery within 30 days before study entry; or have peripheral neuropathy or neuropathic pain Grade 2 or higher. EFFICACY EVALUTIONS: Measurements of M-protein will be followed in serum and 24-hour urine at baseline (prior to treatment on Day 1 of Cycle 1), prior to treatment on Day 1 of Cycles 2-9, and at the Final Visit. The Final Visit/Early Termination Visit will occur 30-42 days after the last dose of Bortezomib. It is recommended that patients who have 100% disappearance of the original monoclonal protein from serum and urine will have the result confirmed by immunofixation. Investigators will also be asked to complete a CRF follow-up form every 6 months for up to 2 years after the Final/Early Termination Visit to capture TTP.

SAFETY EVALUATIONS: A physical examination (including neurological/peripheral neurological examination, vital signs, blood pressure, pulse, respiratory rate, and temperature), karnofsky performance status, hematology, and clinical chemistry tests will be obtained at screening; on Day 1 of each cycle prior to dosing with Bortezomib; and at the Final Visit/Early Termination Visit to occur 30-42 days after the last dose of Bortezomib is administered. Hematology tests will also be obtained prior to dosing during cycles 1 and 2 and every week thereafter. Safety will also be assessed by the reporting of adverse events starting with the signing of the ICF, during treatment, and until the last study related procedure at the Final Visit/Early Termination Visit. The intensity (severity) of the adverse events will be assessed using National Cancer Institute (NCI) common toxicity criteria (CTC) Version 3.0. All adverse events (excluding grade 1 and 2 lab abnormalities) starting with the signing of the ICF, during and until the Final Visit/Early Termination Visit will be recorded on the case report forms (CRFs). Clinically relevant changes in laboratory safety tests, vital signs, and physical/neurological examinations will be recorded as adverse events. Serious adverse events will be reported within 24 hours of knowledge of the event by any member of the investigational site to the sponsor by facsimile (fax), using an SAE form, which will be provided by the sponsor.

STUDY ANALYSIS: Adverse events, serious adverse events, M-protein, extramedullary plasmacytoma measurements, FACT/GOG-Ntx and Karnofsky performance status data will be summarized. Response to study treatment based on M-protein and extramedullary plasmacytoma reduction will also be assessed in the analysis. Patients will receive BMP treatment, consisting of Bortezomib IV bolus infusion 1.3m^2 (twice weekly [Days 1, 4, 8, 11, 22, 25, 29 and 32] for four 6-week cycles [8 doses per cycle]) followed by once weekly [Days 1, 8, 22, and 29] for five 6-week cycles [4 doses per cycle]) in combination with oral melphalan 9mg/m^2 and oral prednisone 60 mg/m^2 once daily on Days 1 to 4 of each 6-week cycle. The max total treatment duration of the study is 54-weeks (9 six-week cycles).

ELIGIBILITY:
Inclusion Criteria:

* Patient is not a candidate for high-dose chemotherapy with stem cell transplant because of age of patient is 65 years or older, overall response in patients less than 65 years old -presence of important comorbid condition(s) likely to have a negative impact on tolerability of high-dose chemotherapy with stem cell transplantation. Sponsor review of these comorbid conditions and approval is required before enrollment
* Symptomatic multiple myeloma or asymptomatic multiple myeloma with related organ or tissue damage
* Presence of measurable disease (secretory multiple myeloma or oligosecretory or nonsecretory multiple myeloma)
* If female, the patient is either postmenopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) from Screening through the Final Visit
* If male, the patient agrees to use an acceptable barrier method for contraception from screening through the Final Visit
* Patient has a Karnofsky performance status >60
* The subject meets the following pretreatment laboratory criteria at and within 14 days before baseline (Day 1 of Cycle 1, before study drug administration): a. platelet count > = 100 x 10^9/L, or > = 70 x 10^9/L if thrombocytopenia is considered by the investigator to be due to myeloma infiltration of bone marrow. b. hemoglobin > = 80 g/L ( > = 4.96 mmol/L) (prior RBC transfusion or recombinant human erythropoietin use is allowed). c. absolute neutrophil count (ANC) > = 1.0 x 10^9/L. d. aspartate aminotransferase (AST) < = 2.5 times the upper limit of normal. e. alanine aminotransferase (ALT) < = 2.5 times the upper limit of normal. f. serum creatinine < = 2 mg/dL (= 176.8 mcmol/L). g. corrected serum calcium < 14 mg/dL ( < 3.5 mmol/L)

Exclusion Criteria:

* Diagnosis of smoldering multiple myeloma or monoclonal gammopathy of undetermined significance (MGUS)
* Diagnosis of Waldenström's disease or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Prior or current systemic therapy for multiple myeloma including steroids (with exception of emergency use of a short course [maximum 4 days] of steroids before randomization or of prior or current use of bisphosphonates)
* Radiation therapy within 30 days before enrollment
* Plasmapheresis within 30 days before enrollment
* Major surgery within 30 days before enrollment (Kyphoplasty is not considered major surgery)
* Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 3.0
* Acute diffuse infiltrative pulmonary and pericardial disease
* Concurrent medical condition or disease (e.g., active systemic infection, uncontrolled diabetes) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada
Locations (3):
- Canada (3):
  - Burnaby, British Columbia
  - Winnipeg, Manitoba
  - N/a N/a